CLINICAL TRIAL: NCT07387471
Title: A Phase 2 Study of Venetoclax Monotherapy in Japanese Subjects With Relapsed or Refractory Waldenström Macroglobulinemia/Lymphoplasmacytic Lymphoma
Brief Title: Study to Assess Change in Disease Activity of Oral Venetoclax in Adult Participants With Recurring Relapsed or Refractory (R/R) Waldenström Macroglobulinemia (WM)/Lymphoplasmacytic Lymphoma (LPL)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M25-558
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Waldenstrom Macroglobulinemia; Lymphoplasmacytic Lymphoma
Keywords: Waldenstrom Macroglobulinemia; Lymphoplasmacytic Lymphoma; Venetoclax; Venclexta; Cancer
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Neoplasms | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Venetoclax Monotherapy (Experimental): Participants will receive venetoclax at doses ramping up to the target dose, as part of the approximately 28 month study duration.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Oral

SUMMARY:
Lymphoplasmacytic Lymphoma (LPL) is a rare type of low-grade B-cell lymphoma. The purpose of this study is to assess the change in disease activity of adult participants with relapsed or refractory Waldenström macroglobulinemia(WM)/LPL receiving venetoclax.

Venetoclax is being investigated in the treatment of WM/LPL. Participants will receive oral venetoclax at doses ramping up to the target dose, as part of treatment. Approximately 14 adult participants with WM/LPL will be enrolled in the study at approximately 20 sites in Japan.

Participants will receive oral venetoclax at doses ramping up to the target dose. The total study duration is approximately 28 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, and checking for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Waldenström macroglobulinemia(WM) /lymphoplasmacytic lymphoma (LPL) according to the 5th edition of the World Health Organization (WHO) classification and/or documented clinicopathological diagnosis of WM in accordance with the consensus panel of the second International Workshop on WM (IWWM).
* At least one prior standard therapy for WM/LPL.
* Measurable disease, defined as follows:

  * WM type LPL population: Immunoglobulin M (IgM) >= 500 mg/dL per central laboratory (approximately 14 participants)
  * Non-IgM type LPL population or IgM < 500 mg/dL: A measurable node having a longest diameter (LDi) greater than 1.5 cm, or a measurable extranodal disease having a LDi greater than 1.0 cm, according to contrast-enhanced computed tomography (CT) scan. (up to 2 participants)
* Requires systemic anti-cancer treatment for WM/LPL, according to the investigator.
* Eastern Cooperative Oncology Group Performance Status < = 2
* Adequate organ and bone marrow function

Exclusion Criteria:

* History of prior exposure to venetoclax or BCL-2 targeted therapy.
* Uncontrolled active systemic infection.
* Known bleeding disorders (e.g., von Willebrand's disease or hemophilia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-03-23 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Major Response | Up to Approximately 28 Months
  Major response is defined as participants with a best overall response of complete response (CR), very good partial response (VGPR) or partial response (PR) per independent review committee (IRC) assessment according to International Workshop on Waldenstrom macroglobulinemia (WM) (IWWM)-11 criteria in participants with Immunoglobulin M (IgM) >= 500 mg/dL at screening.
Number of Participants with Major Response in participants with IgM >= 500 mg/dL | Up to Approximately 28 Months
  Major response is defined as participants with a best overall response of CR, VGPR or PR per IRC assessment according to IWWM-11.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to Approximately 28 Months
  PFS is defined as time from first study treatment to a documented disease progression (PD) according to IWWM-11 criteria, determined by investigator or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to Approximately 28 Months
  OS is defined as time from first study treatment to death due to any cause.
Overall Response (OR) | Up to Approximately 28 Months
  For participants with IgM >= 500 mg/dL at screening, overall response is defined as participants with a best overall response of CR, VGPR, PR or minor response (MR) per investigator assessment according to IWWM-11 criteria. For participants with IgM < 500 mg/dL at screening, overall response is defined as participants with the best overall response of CR or PR per investigator assessment according to Revised Response Criteria for Malignant Lymphoma.
Duration of Response (DOR) | Up to Approximately 28 Months
  For participants with IgM >= 500 mg/dL at screening, DOR is defined as time from the initial response of CR, VGPR or PR per investigator review according to IWWM-11 criteria to PD or death of any cause, whichever occurs first. For participants with IgM < 500 mg/dL at screening, DOR is defined as time from the initial response of CR or PR per investigator review according to Revised Response Criteria for Malignant Lymphoma to PD or death of any cause, whichever occurs first. DOR will be summarized for the participants achieving overall response.
Time to Next Treatment (TTNT) | Up to Approximately 28 Months
  TTNT is defined as time from first study treatment to the starting date of new anti-cancer therapy.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-558